CLINICAL TRIAL: NCT06448481
Title: Aesthetic Outcome of Intra-dermal Versus Transcutaneous Purse-string Closure: a Randomized Evaluator-blinded Split-wound Comparative Effectiveness Trial
Brief Title: Aesthetic Outcome of Intra-dermal Versus Transcutaneous Purse-string Closure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2136552
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Scarring
Keywords: Purse-string
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two blinded observers will record their scores independently using the POSAS instrument.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-dermal purse-string closure on Side A (Experimental): For all participants, one wound side half will be labeled as A and the other side as B. Side A will be closed with a intra-dermal purse-string closure, and Side B will be closed with a transcutaneous purse-string closure.
  Interventions: Procedure: Intra-dermal purse-string closure; Procedure: Transcutaneous purse-string closure
- Intra-dermal purse-string closure on Side B (Experimental): For all participants, one wound side half will be labeled as A and the other side as B. Side B will be closed with a intra-dermal purse-string closure, and Side A will be closed with a transcutaneous purse-string closure.
  Interventions: Procedure: Intra-dermal purse-string closure; Procedure: Transcutaneous purse-string closure

INTERVENTIONS:
Procedure: Intra-dermal purse-string closure — Sutures are placed below the skin surface around a circular surgical wound, and the ends are cinched together like a coin purse.
Procedure: Transcutaneous purse-string closure — Sutures are placed through the skin surface around a circular surgical wound, and cinched together like a coin purse.

SUMMARY:
The purpose of this study is to determine whether intra-dermal versus transcutaneous purse-string closures have similar scar cosmesis and post-operative complications. The investigators will use a split wound model, where half of the wound will be closed with intra-dermal purse-string sutures and the other half will be closed with a transcutaneous purse-string sutures. Three-months post-surgery, the scar will be evaluated via the patient observer scar assessment scale (POSAS), a validated scar instrument, as well as the trace-to-tape method, an objective outcome measure for linear postoperative scars. Any adverse events will also be recorded.

DETAILED DESCRIPTION:
The purse-string closure is a versatile technique that utilizes circumferential tissue advancement for partial or complete closure of circular cutaneous surgical defects. First reported in the 1950s for closure of a malar defect, the purse-string closure is now routinely used for umbilical, urethral, and breast defects as well as for cutaneous surgical defects either alone or in conjunction with top sutures, local flaps, or grafts.

Though the purse-string closure was initially described with circumferentially placed intradermal sutures, various modifications to this technique have been published including sub-cuticular, intra-dermal, and cuticular variations. All modifications of the purse-string closure share the advantages of reduced operating time, decreased defect and scar size, no removal of normal tissue, low hematoma risk, and faster healing time. However, several papers suggest that cuticular (transcutaneous) purse-string closures may be superior to intra-dermal purse-string closures due to enhanced hemostasis from greater compression of the dermal vessels, greater utility in atrophic and actinically damaged skin, lower risk of dermal dehiscence, and better efficacy in skin with limited laxity.

In 2015, a randomized trial comparing secondary intention healing to intradermal purse-string closure found similar cosmetic outcomes, scar size and pain level between the intra-dermal purse-string closure and secondary intention healing however similar studies comparing intra-dermal and transcutaneous purse-string closures are lacking. Given the potential functional advantages of the transcutaneous purse-string closure over the intra-dermal purse-string closure, additional studies comparing the two variations of the purse-string closure are needed to guide clinical practice.

The aesthetic outcome and rate of post-operative complications of intra-dermal versus transcutaneous purse-string closures have not been studied. This study seeks to compare the effectiveness of transcutaneous purse-string sutures to intra-dermal purse-string sutures by using individuals as their own controls in a split-scar model.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure on the head, neck, trunk, or extremities with predicted purse-string closure.
* Willing to return for follow up visit

Exclusion Criteria:

* Incarceration
* Under 18 years of age
* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Observer Scar Assessment as measured by Patient Observer Scar Assessment Score (POSAS) | 3 months
  The primary endpoint will be the score of two blinded reviewers independently using the POSAS assessment. The observer scale of the POSAS consists of six items (vascularity, pigmentation, thickness, relief, pliability, and surface area). All items are scored on a scale ranging from 1 ("like normal skin") to 10 ("worst scar imaginable"). The sum of the six items results in a total score of the POSAS observer scale. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10. All parameters should preferably be compared to normal skin on a comparable anatomic location.

SECONDARY OUTCOMES:
Patient Scar Assessment as measured by Patient Observer Scar Assessment Score (POSAS) | 3 months
  This is the patient portion of the POSAS assessment, which will be independently recorded. The patient scale of the POSAS consists of six items (pain, itch, thickness, color, stiffness, and irregularity). All items are scored on a scale ranging from 1 ("as normal skin") to 10 ("yes, very different"). The sum of the six items results in a total score of the POSAS patient scale. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10.
Width of Scar as measured using Trace-to-Tape Method | 3 months
  The trace-to-tape method is an objective measure for linear postoperative scars. The mean scar width will be determined using the trace-to-tape method. The surface area of the scar will be collected by tracing the scar with a water-based gel pen. While still wet, the gel residue will be lifted from the skin with clear packing tape and transferred on a sheet of paper.
Complications or Adverse Events from Treatment | 3 months
  For example, if one half of the scar has more associated erythema, as measured using the Trace-to-Tape method, then it will be recorded. Other complications from the treatment will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, MD, Principal Investigator — University of California, Davis - Dermatology
Locations (1):
- University of California, Davis - Dermatology Department, Sacramento, California, United States

REFERENCES:
- [Background] Joo J, Custis T, Armstrong AW, King TH, Omlin K, Kappel ST, Eisen DB. Purse-string suture vs second intention healing: results of a randomized, blind clinical trial. JAMA Dermatol. 2015 Mar;151(3):265-70. doi: 10.1001/jamadermatol.2014.2313. PMID 25372450
- [Background] Scholl L, Meier NM, Hessam S, Valavanis K, Bechara FG. Subcuticular and cuticular purse-string sutures in dermatologic surgery. J Dtsch Dermatol Ges. 2016 Feb;14(2):196-8. doi: 10.1111/ddg.12896. Epub 2016 Jan 20. No abstract available. PMID 26788857
- [Background] Fioramonti P, Sorvillo V, Maruccia M, Lo Torto F, Marcasciano M, Ribuffo D, Cigna E. New application of purse string suture in skin cancer surgery. Int Wound J. 2018 Dec;15(6):893-899. doi: 10.1111/iwj.12941. Epub 2018 Jun 29. PMID 29956469
- [Background] Park S, Oh Y, Lee JW, Choi S, Nam KA, Roh MR, Chung KY. Various Applications of Purse-String Suture and Its Cosmetic Outcome in Cutaneous Surgical Defects. Ann Dermatol. 2023 Apr;35(2):100-106. doi: 10.5021/ad.21.263. PMID 37041703
- [Background] Cohen PR, Martinelli PT, Schulze KE, Nelson BR. The cuticular purse string suture: a modified purse string suture for the partial closure of round postoperative wounds. Int J Dermatol. 2007 Jul;46(7):746-53. doi: 10.1111/j.1365-4632.2007.03253.x. PMID 17614809
- [Background] Cohen PR, Martinelli PT, Schulze KE, Nelson BR. The purse-string suture revisited: a useful technique for the closure of cutaneous surgical wounds. Int J Dermatol. 2007 Apr;46(4):341-7. doi: 10.1111/j.1365-4632.2007.03204.x. PMID 17442069
- [Background] Weisberg NK, Greenbaum SS. Revisiting the purse-string closure: some new methods and modifications. Dermatol Surg. 2003 Jun;29(6):672-6. doi: 10.1046/j.1524-4725.2003.29160.x. PMID 12786718
- [Background] Lam TK, Lowe C, Johnson R, Marquart JD. Secondary Intention Healing and Purse-String Closures. Dermatol Surg. 2015 Oct;41 Suppl 10:S178-86. doi: 10.1097/DSS.0000000000000480. PMID 26418684
- [Background] Raposio E, Antonacci M, Caruana G. A simple technique for the excision of cutaneous carcinoma: the round block purse-string suture. World J Surg Oncol. 2014 Aug 20;12:263. doi: 10.1186/1477-7819-12-263. PMID 25142636